CLINICAL TRIAL: NCT00682266
Title: Reducing Cardiovascular Risk Factors In Overweight Adolescents: Multidisciplinary Treatment and Intensity Controlled Interval Training
Brief Title: High-intensity Exercise Training or Multidisciplinary Treatment in Extremely Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 251076
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Adolescent; Overweight; Exercise; multidisciplinary approach; Oxygen uptake; Flow mediated dilatation; Cardiovascular Risk Factors
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic interval training (Experimental): intensity-controlled interval training
  Interventions: Behavioral: intensity controlled interval training (AIT)
- MTG (Experimental): multidisciplinary approach
  Interventions: Behavioral: Multidisciplinary approach (MTG)

INTERVENTIONS:
Behavioral: intensity controlled interval training (AIT) — 4 x 4 min intervals at 90% of maximal heart rate, each interval separated by 3 min at 70%, twice a week for 3 months
  Arms: Aerobic interval training
Behavioral: Multidisciplinary approach (MTG) — exercise, dietary and psychological advice, twice a month for 12 months
  Arms: MTG

SUMMARY:
The aim of the present study was to determine the effects of a multidisciplinary approach and intensity-controlled interval training on cardiovascular risk factors in overweight adolescents

ELIGIBILITY:
Inclusion Criteria:

* BMI >+ 2SD (age adjusted)
* Fitted for group treatment
* at least one parent attending the treatment

Exclusion Criteria:

* Not able to join treatment
* not able to walk

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2004-02; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Flow mediated Diameter Maximal oxygen uptake BMI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rønnaug Ødegård, Dr.med, Study Director — St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Tjonna AE, Stolen TO, Bye A, Volden M, Slordahl SA, Odegard R, Skogvoll E, Wisloff U. Aerobic interval training reduces cardiovascular risk factors more than a multitreatment approach in overweight adolescents. Clin Sci (Lond). 2009 Feb;116(4):317-26. doi: 10.1042/CS20080249. PMID 18673303